CLINICAL TRIAL: NCT05346367
Title: Improving Therapeutic Ratio With Hypo Fractionated Stereotactic Radiotherapy for Brain Metastases
Acronym: SAFESTEREO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haaglanden Medical Centre (Other)
Responsible Party: Principal Investigator, Jaap Zindler, Principal Investigator, MD, PhD, radiation oncologist, Haaglanden Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-115LR
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Brain Metastases
Keywords: fractionated stereotactic radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRT (stereotactic radiotherapy) (Active Comparator): stereotactic radiotherapy in 1 or 3 fractions of 8 Gy up to 15-24 Gy
  Interventions: Radiation: SRT
- fSRT (hypo fractionated stereotactic radiotherapy) (Experimental): hypo fractionated stereotactic radiotherapy in 5 fractions of 7 Gy up to 35 Gy. Brain stem metastases 5 fractions of 6 Gy up to 30 Gy
  Interventions: Radiation: fSRT

INTERVENTIONS:
Radiation: SRT — SRT
  Arms: SRT (stereotactic radiotherapy)
Radiation: fSRT — fSRT
  Arms: fSRT (hypo fractionated stereotactic radiotherapy)

SUMMARY:
Randomized phase II trial. The study aims to investigate a different and potentially safer radio therapeutic treatment method for brain metastases. The current standard of stereotactic radiotherapy (SRT) in one or three fractions is compared to fractionated stereotactic radiotherapy (fSRT) in five fractions.

DETAILED DESCRIPTION:
Randomized phase II trial. Stereotactic radiotherapy is one of the most frequently chosen treatment options for brain metastases. There are an increasing number of long term survivors. Brain necrosis (e.g. radio necrosis) is the most important long term side effect of the treatment, occurring in up to 40% of patients, dependent on the size of the metastasis and delivered radiotherapy dose. Retrospective studies have shown that the incidence of radio necrosis, as well as local tumor recurrence, can be decreased with a risk difference of around 20% by administrating fractionated stereotactic radiotherapy (fSRT, e.g. five fractions) over single fraction stereotactic radiotherapy, especially in large brain metastases. In this trial, one group is treated with SRT in one or three fractions. The other group is treated with fSRT in five fractions. Survival, toxicity and patient reported quality of life are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* At least one brain metastasis of large cell cancer suitable for SRT
* Karnofsky Performance Status ≥ 70
* Ability to provide written informed consent
* New brain metastases during follow-up after surgery allowed (when outside of resection cavity area)
* New brain metastases during follow-up after previous SRT allowed (when outside of previous irradiation field)

Exclusion Criteria:

* Contra-indication for MRI scan
* Primary tumor of small cell lung cancer, germinoma or lymphoma
* Prior whole brain radiotherapy or SRT on the current target brain metastases (in field re-irradiation)
* Presence of leptomeningeal metastases
* Previous inclusion in the SAFESTEREO study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
radio necrosis or local failure | 2 years after treatment
  Incidence of either radio necrosis or local failure according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM).

SECONDARY OUTCOMES:
Survival | 2 years after treatment
  median survival with Kaplan Meyer analysis
symptomatic radio necrosis (RN) or local failure (LF) | 2 years after treatment
  incidence of RN or LF within 2 years after SRT
salvage treatment | 2 years after treatment
  incidence of salvage treatment within 2 years after SRT
distant brain recurrences | 2 years after treatment
  incidence of distant brain recurrences within 2 years after SRT
Dose dexamethasone | baseline - 2 years after treatment
  Dose dexamethasone in mg per day
Anti-epileptic drug use | baseline - 2 years after treatment
  Anti-epileptic drug use in mg per day
Grade 2 or more toxicity (CTCAE v5.0) | baseline - 2 years after treatment
  incidence of Grade 2 or more toxicity according to CTCAE version 5.0 within 2 years after SRT

CONTACTS AND LOCATIONS:
Overall Officials: Jaap D Zindler, MD, PhD, Principal Investigator — Haaglanden MC
Locations (1):
- Haaglanden Medisch Centrum, Leidschendam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crouzen JA, Petoukhova AL, Broekman MLD, Fiocco M, Fisscher UJ, Franssen JH, Gadellaa-van Hooijdonk CGM, Kerkhof M, Kiderlen M, Mast ME, van Rij CM, Nandoe Tewarie R, van de Sande MAE, van der Toorn PPG, Vlasman R, Vos MJ, van der Voort van Zyp NCMG, Wiggenraad RGJ, Wiltink LM, Zindler JD. SAFESTEREO: phase II randomized trial to compare stereotactic radiosurgery with fractionated stereotactic radiosurgery for brain metastases. BMC Cancer. 2023 Mar 25;23(1):273. doi: 10.1186/s12885-023-10761-1. PMID 36964529

DOCUMENTS (1):
  • Study Protocol (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT05346367/Prot_000.pdf